CLINICAL TRIAL: NCT04613154
Title: Magnesium as an Adjunct for Pain Treatment After Surgery for Thumb Base Arthrosis, a Randomised Controlled Study
Brief Title: Magnesium as an Adjunct for Pain Treatment After Surgery for Thumb Base Arthrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in hospital organisation. A large reduction number of patients undergoing surgery.
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 272919
Record Dates: First submitted 2020-09-24; First posted 2020-11-03 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Closed envelope randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Active Comparator): Given 1000 mg oral magnesiumcitrate once daily (4*250mg) during the day of surgery and the next 6 Days.
  Interventions: Dietary Supplement: magnesiumcitrate
- Placebo (Placebo Comparator): Given placebo once daily during the day of surgery and the next 6 Days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: magnesiumcitrate — Magnesiumcitrate 250 mg, Apoteket AB, Sweden
  Arms: Magnesium
Dietary Supplement: Placebo — Ester-c
  Arms: Placebo

SUMMARY:
A randomised controlled trial of addition to the standard pain treatment of 1000 mg oral magnesium citrate or placebo for 7 Days during surgery for thumb base arthrosis. Intraoperative nociception will be measured with the NoL-index with a PM-200 machine.

DETAILED DESCRIPTION:
Our hypothesis is that an addition of oral 1000 mg magnesium citrate daily for 7 Days starting at the day of the surgery will decrease the postoperative pain and improve the recovery after surgery. It will be given as an supplement to the regular pain treatment with acetaminophen and oxycodone that are used in our hospital and compared to a placebo. The choice of treatment will be blinded for the patient, the care providers and for the research team doing the evaluation.

The pain level will be collected Before surgery, postoperatively and at 14 Days after surgery and by a self reporting form during the first 7 Days. The patients will also report their recovery with a modified QoR-15 form. QoR-15 is validated in a Swedish version.

Magnesium is shown to reduce postoperative pain in some studies that used iv magnesium sulphate. For long lasting pain conditions oral magnesium is shown to improve the patients well being and decrease their pain in some conditions. Magnesium acts as a mild antagonist at the NMDA-receptor. Thus low levels of magnesium is thought to increase the risk of long lasting postoperative pain. Therefore there are reason to expect a higher dose of magnesium supplement decreases the long lasting post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Planned for surgery of thumb base arthrosis with trapeziectomy with ligament reconstruction tendon interposition.
* Age 18 years or older.
* low anesthetic risk, ASA class 1 or 2.
* Be able to take oral medication.
* Be able to read and communicate in Swedish.

Exclusion Criteria:

* Age under 18 years.
* Heartfailure, kidney failure, ischemic hearth disease.
* Previous neuropathic pain or complex pain syndrome.
* Serious psychiatric morbidity
* Not able to communicate in Swedish
* Skin problems that makes the application of NoL-sensor impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Pain after 48 hours from surgery | Self reported at 48 hours after surgery.
  Pain measured with a self reported written numerical rating scale with eleven steps 0-10 where 0 is no pain and 11 is the worst pain possible (NRS) after 48 h after surgery.

SECONDARY OUTCOMES:
QoR15swe (Quality of Recovery, a 15 item questionaire translated to swedish) | Day 1 to day 7 after surgery.
  Recovery measured by QoR15swe day 1-7. A written form filled in by the patients and returned to the hospital by mail. QoR15 is a recovery score with 15 items that gives a score between 0-150. 0 points indicates worst possible recovery and 150 indicates best possible recovery. We are using a swedish translation validated by Lyckner et al 2018.
Pain 1 hour after surgery | 1 hour after leaving the operating theatre
  Pain measured with an oral numerical rating scale with eleven steps 0-10 where 0 is no pain and 11 is the worst pain possible (NRS) reported to the staff at the post operative ward 1 hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Pether Jildenstål, phd, Principal Investigator — Universitetssjukhuset Örebro, ANIVA-kliniken
Locations (1):
- Örebro University Hospital, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Shin HJ, Na HS, Do SH. Magnesium and Pain. Nutrients. 2020 Jul 23;12(8):2184. doi: 10.3390/nu12082184. PMID 32718032
- [Background] Cowen R, Stasiowska MK, Laycock H, Bantel C. Assessing pain objectively: the use of physiological markers. Anaesthesia. 2015 Jul;70(7):828-47. doi: 10.1111/anae.13018. Epub 2015 Mar 14. PMID 25772783
- [Background] Brown EN, Pavone KJ, Naranjo M. Multimodal General Anesthesia: Theory and Practice. Anesth Analg. 2018 Nov;127(5):1246-1258. doi: 10.1213/ANE.0000000000003668. PMID 30252709
- [Background] Lyckner S, Boregard IL, Zetterlund EL, Chew MS. Validation of the Swedish version of Quality of Recovery score -15: a multicentre, cohort study. Acta Anaesthesiol Scand. 2018 Aug;62(7):893-902. doi: 10.1111/aas.13086. Epub 2018 Feb 7. PMID 29417552
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Yousef AA, Al-deeb AE. A double-blinded randomised controlled study of the value of sequential intravenous and oral magnesium therapy in patients with chronic low back pain with a neuropathic component. Anaesthesia. 2013 Mar;68(3):260-6. doi: 10.1111/anae.12107. Epub 2012 Dec 17. PMID 23384256